CLINICAL TRIAL: NCT00898183
Title: Cytogenetic, Molecular and Cellular Biology Studies in Metastatic Melanoma Patients, Ancillary
Brief Title: S9431: Studying Genes and Immune Response in Tumor Samples From Patients With Locally Advanced or Metastatic Melanoma
Status: Completed | Type: Observational
Sponsor: SWOG Cancer Research Network (Network)
Collaborators: National Cancer Institute (NCI) (NIH); Eastern Cooperative Oncology Group (Network)
Responsible Party: Sponsor
Other Study IDs: CDR0000078645; SWOG-9431 (Other: SWOG); U10CA032102 (NIH)
Record Dates: First submitted 2009-05-09; First posted 2009-05-12 (Estimated); Last update posted 2018-06-28 (Actual); Status verified 2013-02

CONDITIONS: Melanoma (Skin)
Keywords: stage III melanoma; stage IV melanoma; recurrent melanoma
MeSH Terms: conditions — Melanoma | interventions — Gene Expression Profiling; Amplified Fragment Length Polymorphism Analysis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Genetic: gene expression analysis
Genetic: polymorphism analysis

SUMMARY:
RATIONALE: Studying samples of tumor tissue and blood from patients with cancer in the laboratory may help doctors learn more about changes that occur in DNA and identify biomarkers related to cancer. It may also help doctors predict how patients will respond to treatment.

PURPOSE: This laboratory study is assessing genes and immune response in tumor samples from patients with locally advanced or metastatic melanoma.

DETAILED DESCRIPTION:
OBJECTIVES:

* Characterize the frequency of non-random cytogenetic abnormalities in regional and distant melanoma metastases and explore their association with clinical outcome of patients with metastatic melanoma.
* Characterize the frequency of specific genetic alterations at either the DNA, mRNA, or protein level and explore the association of these abnormalities with clinical outcome in these patients.
* Characterize the host immunologic response to metastatic melanoma by determining whether the in vivo pattern of cytokine expression is consistent with specific subsets of T helper cells within melanoma deposits and to explore whether host immunologic response varies based on the site of metastatic disease and/or correlates with clinical outcome in these patients.
* Obtain peripheral blood, sera, and paraffin embedded tumor blocks from these patients.
* Correlate the most prevalent gene copy alteration observed in metastatic disease with the risk of progression in tissue samples from patients registered on SWOG-9035 (primary melanoma).

OUTLINE: Fresh and snap frozen tumor tissue samples are obtained from biopsy or surgical procedures in the coordinated study. Specimens undergo mRNA and DNA analysis of tumor-related genes and cytokine gene expression. Peripheral blood samples are obtained and processed for sera and mononuclear cell testing. Tumor tissue samples embedded in paraffin or on unstained slides are also obtained.

PROJECTED ACCRUAL: Approximately 120 patients will be accrued for this study within 3-4 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of stage III or IV metastatic melanoma

  * Concurrent enrollment on a SWOG-coordinated melanoma treatment study (within 56 days of registration on this study) OR
  * Previously enrolled on and eligible for at least 1 SWOG-coordinated melanoma study and scheduled to undergo biopsy/surgery for regional lymph node or disseminated metastatic disease OR
  * Concurrent enrollment on SWOG-9430 (FISH analysis)

PATIENT CHARACTERISTICS:

Age

* Not specified

Performance status

* Not specified

Life expectancy

* Not specified

Hematopoietic

* Not specified

Hepatic

* Not specified

Renal

* Not specified

PRIOR CONCURRENT THERAPY:

Biologic therapy

* Not specified

Chemotherapy

* Not specified

Endocrine therapy

* Not specified

Radiotherapy

* Not specified

Surgery

* Not specified

Other

* Not previously enrolled on SWOG-9431

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 91 (Actual)
Dates: Start 1996-11; Primary Completion 2006-02 (Actual); Study Completion 2007-02 (Actual)

PRIMARY OUTCOMES:
Correlation of frequency of non-random cytogenetic abnormalities in regional and distant melanoma metastases with clinical outcome
Correlation of frequency of specific genetic alterations at either the DNA, mRNA, or protein level with clinical outcome
Host immunologic response to metastatic melanoma (i.e., in vivo pattern of cytokine expression consistent with specific subsets of T helper cells within melanoma deposits)
Variation and correlation of host immunologic response with site of metastatic disease and/or clinical outcome
Development of a tissue bank (peripheral blood, sera, and paraffin-embedded tumor blocks)
Correlation of the most prevalent gene copy alteration observed in metastatic disease with the risk of progression

CONTACTS AND LOCATIONS:
Overall Officials: David M. Gustin, MD, Study Chair — University of Chicago; John M. Kirkwood, MD, Study Chair — University of Pittsburgh

REFERENCES:
- [Result] Moore SR, Persons DL, Sosman JA, Bobadilla D, Bedell V, Smith DD, Wolman SR, Tuthill RJ, Moon J, Sondak VK, Slovak ML. Detection of copy number alterations in metastatic melanoma by a DNA fluorescence in situ hybridization probe panel and array comparative genomic hybridization: a southwest oncology group study (S9431). Clin Cancer Res. 2008 May 15;14(10):2927-35. doi: 10.1158/1078-0432.CCR-07-4068. PMID 18483359